CLINICAL TRIAL: NCT06777394
Title: Effects of High Intensity Interval Training on Endurance and Trunk Stability in Children With Down Syndrome
Brief Title: Effects of High Intensity Interval Training in Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0718
Record Dates: First submitted 2024-11-03; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Down Syndrome
Keywords: Down Syndrome,.; High intensity interval training; Endurance; Trunk Stability
MeSH Terms: conditions — Down Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment it will be randomized control trail in which non probability convenient sampling will be used . Two groups of 3-14 age will be formed in which participants will be randomly divided. Group A will be receive Group Task- Oriented Training. Group B wil be receive routine therapy
Who Masked: Participant
Masking Description: Single (Participants) Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): task oriented training, group A perform high intensity interval training in addition to routine physical therapy routine exercise giving short burst of intense work for 15 second to 4 mins
  Interventions: Other: High intensity interval training
- control group (Other): Routine treatment , streching and normal range of motion exercise should be taught to the patients. low intensity and aerobic exercise perform
  Interventions: Other: Routine treatmet

INTERVENTIONS:
Other: High intensity interval training — The HIIT program begins with a warm-up, followed by high-intensity repetitions separated by moderate-intensity recovery intervals. High-intensity exercises are performed near maximum effort, while moderate-intensity periods are maintained at 50% effort. HIIT exercises, involving low-skill movements in short bursts, enhance blood sugar regulation and fat-burning capacity.
  The HIIT protocol has four phases:
  Warm-Up: 10 minutes, gradually increasing to about 60% of maximum heart rate. Intervals: 4 minutes at 85-95% maximum heart rate. Relief/Recovery: 3 minutes at 60% maximum heart rate, repeated four times. Cool Down: 5 minutes, bringing the heart rate down to around 50% of maximum. Three key components determine the success of HIIT: intensity, duration, and recovery period. Exercises include dumbbell and kettlebell exercises, push-ups, squats, jump training, and stationary cycling
  Arms: Experimental group
Other: Routine treatmet — outine physical therapy includes stretching exercises, exercises to maintain a normal range of motion, and low-intensity and aerobic exercises for the patients.
  Low-Intensity Exercise: The effects of low-intensity exercise become noticeable after about 20 minutes, providing a metabolic boost during the activity. Generally, a longer exercise duration further enhances metabolism.
  Arms: control group

SUMMARY:
Down Syndrome (DS), a genetic condition marked by the presence of an extra chromosome 21, is associated with various cognitive and physical challenges. Children with DS often experience motor development issues, including reduced endurance and decreased trunk stability, which underscores the need for targeted interventions. Common impairments in individuals with DS include hypotonia, ligament laxity, reduced muscle strength, limited muscle co-contraction, poor postural control, and impaired proprioception. This study is driven by a lack of research on the effects of High-Intensity Interval Training (HIIT) in this population, despite its documented benefits in enhancing cardiovascular fitness across other groups. Existing literature supports the benefits of exercise interventions for people with DS, but the application and advantages of HIIT-particularly concerning endurance and trunk stability-are underexplored.

DETAILED DESCRIPTION:
The study aims to evaluate the impact of a structured HIIT program on endurance and trunk stability in children with DS. Conducted as a randomized controlled trial (RCT) at Khuwaja Arshad Hospital, Sargodha, the study will include 30 participants divided equally and randomly assigned to two groups. The inclusion criteria include children with a confirmed DS diagnosis, aged 3 to 14, with the ability to understand instructions, stand, and walk independently, and of any gender. Exclusion criteria include mobility impairments, signs of atlantoaxial joint instability, and neurological conditions. Group A will participate in a HIIT program, while Group B will receive routine physical therapy. Pre- and post-intervention assessments will use validated tools to measure endurance (6-Minute Walk Test) and trunk stability (Functional Reach Test). Additionally, the feasibility and acceptability of the HIIT program will be qualitatively evaluated. Data will be collected at baseline and post-intervention and analyzed using SPSS version 23.Data analysis will be conducted using SPSS software. Quantitative data will be reported as mean and standard deviation and visualized with histograms, while qualitative data will be summarized as frequency and percentage and displayed using bar charts. Statistical techniques will be applied to compare baseline characteristics between groups and to assess normal distribution through the Four Square Step Test, the Six-Minute Walk Test for endurance, and the Functional Reach Test for trunk stability. If data follow a normal distribution, within-group differences will be analyzed using a paired sample t-test; otherwise, the Wilcoxon Signed Rank test, a non-parametric alternative, will be applied. For between-group differences, an independent sample t-test will be used for normally distributed data, while the Mann-Whitney U test will be used for non-normally distributed data. A 95% confidence interval and a significance level of p < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 3 to 14 years
* clinically diagnose in children with down syndrome

Exclusion criteria

* Any neurological condition
* History of dementia

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Four square balance test | 6 weeks
  a tool having dynamic balance and coordination. its ability to step over low objects, forward , sideways and backward

SECONDARY OUTCOMES:
6 minutes walk test for endurance | 6 weeks
  A tool used to monitor response to treatments for heart lungs and other health problem for simple measure of functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Sheza Khan, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonarakis SE, Skotko BG, Rafii MS, Strydom A, Pape SE, Bianchi DW, Sherman SL, Reeves RH. Down syndrome. Nat Rev Dis Primers. 2020 Feb 6;6(1):9. doi: 10.1038/s41572-019-0143-7. PMID 32029743